CLINICAL TRIAL: NCT01612663
Title: Comparison of Different Acupuncture Methods on Knee Pain
Brief Title: Effect of Distal Needling on Knee Pain Using Acupuncture Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Elyad Davidson, PI Head Pain Unit, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 007212-HNO-CTIL
Record Dates: First submitted 2012-06-03; First posted 2012-06-06 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Patellar Tendonitis; Complete Tear, Knee, Anterior Cruciate Ligament
Keywords: Knee pain; Acupuncture; Sham acupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- deep needle non-site specific (Active Comparator)
  Interventions: Device: Pain relief by Acupuncture needle at non-specific site
- contralateral elbow to the knee pain (Active Comparator)
  Interventions: Device: Acupuncture needle
- Energy of Living Systems Needling (Active Comparator)
  Interventions: Device: Acupuncture needle
- Sham acupuncture (Placebo Comparator)
  Interventions: Device: Acupuncture needle

INTERVENTIONS:
Device: Pain relief by Acupuncture needle at non-specific site
  Arms: deep needle non-site specific
Device: Acupuncture needle
  Arms: contralateral elbow to the knee pain
Device: Acupuncture needle
  Arms: Energy of Living Systems Needling
Device: Acupuncture needle
  Arms: Sham acupuncture

SUMMARY:
The purpose of this study is to test if specific therapeutic benefits of acupuncture are mostly attributable to contextual and psychosocial factors, such as patients' beliefs and expectations.The investigators propose using the 2 acupuncture methods, which refrains from inserting needles in the affected area, in order to evaluate the short-term and long-term efficacy of acupuncture in a clinical setting compared with placebo and compared with invasive needling that does not adhere to "correct" acupuncture rules.

DETAILED DESCRIPTION:
The main novel features of this study:

1. First aim to assess the effect of distal needling on knee pain
2. Second aim to directly compare two acupuncture techniques, placebo, needling at "wrong" places and "correct" needling for knee pain

Advantages of the study compared to published data:

1. Distal needling - enables assessment of range of motion (ROM) and pain level during needling.
2. Both acupuncture systems rely on minimal questioning, which simplifies the patient-practitioner interactions.
3. Exploratory studies in the clinic of DP show that it is possible to distinguish between "correct" and "incorrect" needling, at least in the short term. Long term effects have not been assessed yet.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old), suffering chronic stable pain score >40 mm on 100 mm VAS of the knee due to patellar tendonitis.
* Patients have had X-rays or other tests confirming they are not candidates for surgery nor are scheduled for steroid injections or hyaluronic acid injections within 8 weeks from the beginning of the study.
* Adult patients (> 18 years old), two weeks after ACL reconstruction surgery (with or without meniscal involvement), with pain score >40 mm on 100 mm VAS of the knee (all patients at this stage have significant ROM limitation).

Exclusion Criteria:

* Patient refusal
* Soldiers
* Pregnancy
* Morbid obesity
* Diabetes
* Peripheral vascular disease
* Lower limb neurological deficit (such as multiple sclerosis, nerve palsy), other serious co-morbidity (including severe back pain or hip pain)
* A history of prolonged or current steroid use
* Received hyaluronic acid injections within the previous 3 months
* Have needle phobia or allergy to sticking plaster.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Effect of Distal Needling on Knee Pain Using Acupuncture Techniques | 2 years
  Effect of Distal Needling on Knee Pain Using 4 different Acupuncture Techniques by:
  1. Pain measurement by Visual Analogue Scale (VAS)
  2. Range of motion (ROM)

CONTACTS AND LOCATIONS:
Overall Officials: Elyad Davidson, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Please Select, Israel